CLINICAL TRIAL: NCT06800404
Title: "A Phase 2, Open Label, Efficacy and Safety Study of Autologous HB-adMSCs for the Treatment of Patients With Multiple Sclerosis"
Brief Title: "HB-adMSCs for the Treatment of Patients With Multiple Sclerosis"
Acronym: MS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBMS02
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS); Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Stem Cells; Hope Biosciences; MS; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Autologous adipose-derived HB-adMSCs
  Interventions: Drug: Autologous HB-adMSCs

INTERVENTIONS:
Drug: Autologous HB-adMSCs — Autologous HB-adMSCs

SUMMARY:
This protocol is part of a clinical study to evaluate efficacy and safety of multiple intravenous administrations of HB-adMSCs for the treatment of Multiple Sclerosis.

DETAILED DESCRIPTION:
This clinical trial is designed as an open label, single center, phase 2 study to assess the efficacy and safety of multiple autologous adipose derived mesenchymal stem cells in patients with Relapsing Remitting Multiple Sclerosis. The trial includes a screening period of up to 4 weeks, a 32-week treatment period, and a safety Follow-up period of 20 weeks after the last investigational product administration. This clinical trial will be opened to enroll up to 10 eligible subjects diagnosed with Relapsing Remitting Multiple Sclerosis. Each eligible study subject will receive a total of 6 intravenous infusions of HB-adMSCs. Study infusions will be administered with the following regimen, Week 0, 4, 8, 16, 24 and 32, this dosing interval has been selected because due to the efficacy observed in the completed placebo-controlled counterpart to this study, HBMS01 (IND 027633, NCT05116540). Efficacy was observed at the end of study visit (week 52), post-therapy with six infusions of HB-adMSCs. The following objectives will be investigated: efficacy as determined by the Multiple Sclerosis Quality of Life (MSQOL-54) Instrument, efficacy as determined by changes in Expanded Disability Status Scale (EDSS), safety as determined by changes in Patient Health Questionnaire (PHQ-9), and safety as determined by the incidence of adverse events or serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 - 75 years of age.
2. Study subjects must have been diagnosed with Relapsing Remitting Multiple Sclerosis (RRMS) for at least 6 months before study participation.
3. Study subjects must have been randomized into the placebo group and completed participation in the HBMS01 clinical trial (IND 027633). (A randomized, double-blind, single center, phase 2 clinical trial that assessed the efficacy and safety of autologous HB-adMSCs vs placebo for the treatment of patients with Multiple Sclerosis.)
4. Study subjects must be stabilized on any MS therapy for at least 6 months prior to enrollment.
5. Study subjects must agree not to increase or begin any Diseases Modifying Therapies for MS during participation in the clinical trial.
6. Study subjects must have an EDSS score between 3.0 to 6.5. (Patient must be able to walk).
7. Study subjects must have previously banked their mesenchymal stem cells with Hope Biosciences.
8. Study subjects should be able to read, understand and to provide written consent.
9. Before any clinical-trial-related procedures are performed, informed consent must be obtained from the subjects voluntarily.
10. Female study subjects of childbearing potential should not be pregnant or plan to become pregnant during study participation and for 6 months after the last investigational product administration. Female study subjects of childbearing potential should confirm the use of one of the following contraceptive measures:

    * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
    * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
    * Barrier contraceptive methods (condoms, diaphragm, etc.).
    * Surgery (occlusion bilateral tubal ligation, hysterectomy, vasectomized partner).
11. Male subjects if their sexual partners can become pregnant should ensure the use one of the following methods of contraception during study participation and for 6 months after the last administration of the investigated product:

    * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
    * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
    * Barrier contraceptive methods (condoms, diaphragm, etc.).
    * Surgery (vasectomy, occlusion bilateral tubal ligation (partner), hysterectomy (partner)).
12. Study subject is able and willing to comply with the requirements of this clinical trial.
13. Subjects in the study should have evidence of disease, as shown by MRIs of the brain or spinal cord, with the most recent being within 1 year of the screening date.

Exclusion Criteria:

1. Women who are currently pregnant or lactating.
2. Study subject has any active malignancy, including but not limited to evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
3. Study subject has known addiction or dependency or has current substance use or abuse.
4. Study subject has 1 or more significant concurrent medical conditions (verified by medical records), including the following:

   * Poorly controlled diabetes mellitus (PCDM) defined as history of deficient standard of care treatment and/or pre-prandial glucose >130mg/dl during screening visit or post-prandial glucose >200mg/dl.
   * Medical History of Chronic kidney disease (CKD) diagnosis and/or screening results of eGFR < 59mL/min/1.73m2
   * Presence of New York Heart Association (NYHA) Class III/IV heart failure during screening visit.
   * Any medical history of myocardial infarction in any of the different types, such as ST-elevation myocardial infarction (STEMI) or non-ST-elevated myocardial infarction (NSTEMI), coronary spasm, or unstable angina.
   * Medical history of uncontrolled high blood pressure defined as a deficient standard of care treatment and/or blood pressure > 180/120 mm/Hg during screening visit.
   * Medical history of diseases such as, inherited thrombophilias, cancer of the lung, brain, lymphatic, gynecologic system (ovary or uterus), or gastrointestinal tract (like pancreas or stomach).
   * Medical history of conditions, such as recent major general surgery, (within 12 months before the Screening), lower extremity paralysis due to spinal cord injury, fracture of the pelvis, hips, or femur.
5. Study subject has received any stem cell treatment within 12 months before first dose of investigational product other than stem cells produced by Hope Biosciences.
6. The study subject has received any experimental drug within 12 months before the first dose of the investigational product. (Except for COVID-19 vaccinations)
7. Study subject has a laboratory abnormality during screening, including the following:

   * White blood cell count < 3000/mm3
   * Platelet count < 80,000mm3
   * Absolute neutrophil count < 1500/mm3
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 10 upper limit of normal (ULN) x 1.5
8. Study subject has any other laboratory abnormality or medical condition which, in the opinion of the investigator, poses a safety risk or will prevent the subject from completing the study.
9. The study subject has any concurrent neurologic disease, including hereditary conditions that the principal investigator considers could interfere with the study participation. Some of these neurologic diseases could be Charcot-Marie-Tooth (CMT) or Spinocerebellar Ataxia (SCA).
10. Study subject is unlikely to complete the study or adhere to the study procedures.
11. Study subject has a previously diagnosed psychiatric condition which in the opinion of the investigator may affect self-assessments.
12. Study subject with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days prior to first dose of the investigational product.
13. Male study subjects who plan to donate sperm during the study or within 6 months after the last dose. Female patients who plan to donate eggs or undergo in vitro fertilization treatment during the study or within 6 months after the last dose.
14. Study subjects who are determined by the Investigator to be unsuitable for study enrollment for other reasons.
15. Subjects' life expectancy must not have been considerably limited by other comorbidities, a history of previous myelodysplasia, or hematologic illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Multiple Sclerosis Quality of Life (MSQOL)-54 Instrument scores | 1 year
  The MSQOL-54 is a comprehensive health-related quality of life measure incorporating general and MS-specific questions into a single instrument.
  The developers used the SF-36 as a base and added 18 questions to address MS-specific problems, including fatigue and cognitive function.
  This 54-item questionnaire provides 12 sub-scales, two summary scores, and two extra single-item measures. The sub-scales are physical function, role limits-physical, emotional role restrictions, pain, emotional well-being, energy, health perceptions, social position, cognitive function, health distress, overall quality of life, and sexual function. There is no single overall score for MSQOL-54. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores (scale scores range from 0 to 100 and a higher scale score indicates improved quality of life).

SECONDARY OUTCOMES:
Change from Baseline in Expanded Disability Status Scale (EDSS) scores | 1 year
  The EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. This scale ranges from 0 to 10 in 0.5-unit increments and a higher score represents increased disability. Scoring is based on an examination by a neurologist.
Change from Baseline in Patient Health Questionnaire (PHQ-9) scores | 1 year
  The PHQ-9 is the most used depression and suicidal thoughts screening test used to monitor the severity of depression and response to treatment. Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Incidence of treatment-emergent Adverse Event (TEAEs) | 1 year
  The number of patients and count of TEAEs of all patients in the study
Incidence of serious Adverse Events (SAEs) | 1 year
  Incidence of serious Adverse Events (SAEs)
Incidence of AEs of special interest (serious or nonserious) | 1 year
  Incidence of AEs of special interest (serious or nonserious), including thromboembolic events, peripheral events defined as, thromboembolism of the extremities, also infections and hypersensitivities.
Clinically significant changes in laboratory value results | 1 year
  Clinically significant changes in laboratory values results (laboratory values assessed will be separated into different outcomes by respective unit)
Clinically significant changes in vital signs | 1 year
  Clinically significant changes in vital signs (vital signs assessed will be separated into different outcomes by respective unit)
Clinically significant changes in weight | 1 year
  Clinically significant changes in weight (measured in pounds)
Clinically significant changes in physical examination results | 1 year
  Clinically significant changes in physical examination results
Clinically significant changes in Multiple Sclerosis concomitant medications | 1 year
  Clinically significant changes in Multiple Sclerosis concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Research Foundation
Locations (1):
- Hope Biosciences Research Foundation, Sugar Land, Texas, United States